CLINICAL TRIAL: NCT02446665
Title: Comprehensive Evaluation of Disease Status in Primary Sclerosing Cholangitis by MRCP and MR Elastography Through Hepatic Fibrosis Estimation With Comparison to FibroScan
Brief Title: Disease Status in Primary Sclerosing Cholangitis by Elastography
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-5707
Record Dates: First submitted 2015-02-20; First posted 2015-05-18 (Estimated); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Primary Sclerosing Cholangitis; Elastography; Hepatic Fibrosis; Magnetic Resonance Imaging
MeSH Terms: conditions — Cholangitis, Sclerosing; Liver Cirrhosis | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- PSC Patients (Experimental): MR Elastography, Fibroscan and standard of care biopsy
  Interventions: Device: MR Elastography (MRE) and FibroScan
- Non-PSC Patients (Active Comparator): MR Elastography, Fibroscan and standard of care biopsy
  Interventions: Device: MR Elastography (MRE) and FibroScan

INTERVENTIONS:
Device: MR Elastography (MRE) and FibroScan

SUMMARY:
Primary sclerosing cholangitis (PSC) is a chronic liver disease that can lead to liver cirrhosis, liver failure and liver cancer. Assessment of disease status is important to determine optimal treatment but the diagnosis of PSC is challenging. There is a dire need of an accurate non-invasive tool for longitudinal assessment of PSC. MR Elastography (MRE) has been recently proven to estimate liver fibrosis noninvasively and accurately. Estimation of liver fibrosis by MRE along with imaging derived morphological information (MRCP) will be utilized in this study comprehensively to provide a surrogate non-invasive imaging biomarker for monitoring disease status in PSC. Successful outcomes will provide an opportunity for optimal treatment triage including liver transplantation via accurate and non-invasive estimation of true disease status in PSC.

DETAILED DESCRIPTION:
Primary sclerosing cholangitis (PSC) is a chronic liver disease that causes inflammation and obstruction of bile ducts. It can eventually lead to liver cirrhosis due to fibrosis, liver failure and liver cancer. The diagnosis of PSC is challenging as there is no single diagnostic test and usually involves a multidisciplinary approach with MRI playing a major role. Assessment of disease status is important to triage patients for optimal treatment including liver transplantation and prevention of liver failure. There are however no established blood tests that can reliably track the disease progression and repeated liver biopsies have multiple drawbacks including complications, costs and feasibility. There is a dire need of an accurate non-invasive tool for longitudinal assessment of PSC. MR Elastography (MRE) has been recently proven to estimate liver fibrosis noninvasively and accurately. Estimation of liver fibrosis by MRE along with imaging derived morphological information (MRCP) will be utilized in this study comprehensively to provide a surrogate non-invasive imaging biomarker for monitoring disease status in PSC. The patients would have or will agree to undergo a liver FibroScan examination to grade fibrosis within 3 months of the MRI examination. In addition to the standard protocol liver and biliary MR examination including MRCP and contrast enhanced imaging, MRE will be added to the study exam following informed consent. A control group of non-PSC subjects with known chronic liver disease such as chronic viral hepatitis who have had liver biopsy and FibroScan within similar time frame of 3 months, to assess fibrosis grade will also undergo MR Elastography in order to validate the results of fibrosis by MRE. The study has significant implications for care of patients with PSC. Successful outcomes will provide an opportunity for optimal treatment triage including liver transplantation via accurate and non-invasive estimation of true disease status in PSC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known PSC
* Control group of patients with Non-PSC chronic liver disease with recent (<3month) liver biopsy and under imaging surveillance.

Exclusion Criteria:

* General Contraindications to MRI such as pacemaker, brain aneurysm clips etc.
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2014-10; Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Validation of fibrosis quantification via MR Elastography | The elastography will be done at the time when the participant would be undergoing their normal clinical care, at the time specified by the primary care physician's order (within 3 months of the MRI examination)

CONTACTS AND LOCATIONS:
Overall Officials: Kartik Jhaveri, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada